CLINICAL TRIAL: NCT05700097
Title: A Phase II, Randomized, Double-blind, Placebo-controlled, Dose-Finding, Multi-center Study to Assess the Efficacy and Safety of Dengzhanxixin Injection in Patients With Acute Ischemic Stroke Receiving Reperfusion Therapy
Brief Title: Dengzhanxixin Injection for Acute Ischemic Stroke Receiving Reperfusion Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCRC-2022-02
Record Dates: First submitted 2022-11-16; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Dose Arm (Experimental): Dengzhanxixin injection 40ml/day, placebo 40ml/day. Dengzhanxixin injection 40ml, diluted with 250ml of 0.9% sodium chloride injection and then slowly intravenously infused once a day; placebo injection 40ml, diluted with 250ml of 0.9% sodium chloride injection and then slowly intravenously infused once a day.
  Interventions: Drug: Dengzhanxixin Injection
- High Dose Arm (Experimental): Dengzhanxixin injection 80ml/day. Dengzhanxixin injection 40ml, diluted with 250ml of 0.9% sodium chloride injection, and then slowly intravenously infused twice a day.
  Interventions: Drug: Dengzhanxixin Injection
- Placebo Arm (Placebo Comparator): Placebo injection 80ml/day. Placebo injection 40ml, diluted with 250ml of 0.9% sodium chloride injection, and then slowly intravenously infused twice a day.
  Interventions: Drug: Placebo injection

INTERVENTIONS:
Drug: Dengzhanxixin Injection — Experimental arms for low, and high dose for the standard protocol
  Other Names: Dengzhanxixin Zhusheye
  Arms: High Dose Arm; Low Dose Arm
Drug: Placebo injection — placebo control arm for the standard protocol
  Other Names: Placebo
  Arms: Placebo Arm

SUMMARY:
To assess the Efficacy and Safety of Dengzhanxixin Injection in Patients With Acute Ischemic Stroke Receiving Reperfusion Therapy.

DETAILED DESCRIPTION:
To evaluate the safety and efficacy of Dengzhanxixin at different doses of 80ml/day, 40 ml/day, or placebo within 24 hours after the onset of ischemic stroke. The primary objective of this study is the proportion of subjects with excellent outcomes defined as mRS (0-1) among the three treatment groups at 90 days.

ELIGIBILITY:
Inclusion Criteria:

* More than or equal to 18 years old and less than 80 years old;
* Acute ischemic stroke confirmed by computed tomography (CT) or magnetic resonance imaging (MRI) of the head;
* Stroke onset within 24 hours and can be treated with study drug within 24 hours of symptoms onset；
* The patient has received or is planning to receive vascular reperfusion therapy after onset；
* Baseline NIHSS score is ≥4 and ≤26.
* mRS ≤1 prior onset.
* Informed consent signed.

Exclusion Criteria:

* Intracranial hemorrhage: cerebral hemorrhage, subarachnoid hemorrhage, etc.;
* The acute infarcts lesion Involvement of more than one-third of middle cerebral artery (MCA) territory on initial brain imaging;
* Rapidly improving symptoms at the discretion of the investigator;
* Patients who have taken Dengzhanxixin Injection，edaravone or other brain protective drugs after onset ;
* History of intracranial hemorrhage；
* History of severe head trauma, stroke or myocardial infarction in past 3 months;
* Diagnosised intracranial tumor and giant intracranial aneurysm；
* Diagnosised aortic arch dissection；
* Undergoing major surgery within 2 weeks prior to screening; or intracranial or intraspinal surgery within 3 months prior to screening;
* Currently accompanied by active visceral bleeding; or arterial puncture at a site that is not easy to compress hemostasis within 1 week before screening; or gastrointestinal or urinary system bleeding occurred within 3 weeks before screening;
* Those with acute bleeding tendency, including: platelet count <100×109/L, combined with hemophilia, etc.; or those with partially activated thrombin time greater than 3 times the upper limit of normal;
* Oral anticoagulants, and international normalized ratio>1.7 or prothrombin time>15s;
* Diagnosed primary liver and kidney disease, AST or ALT (>2 times the ULN), serum creatinine >2.0mg/dL or >176.8µmol/L;
* Persistent blood pressure elevation ( systolic ≥180 mmHg or diastolic ≥100 mmHg ), despite blood pressure lowering treatment;
* Those with a history of epilepsy or epilepsy-like symptoms at the onset of stroke;
* Complete atrioventricular block; or according to the New York Heart Association (NYHA) cardiac function class II or above; or have been hospitalized due to congestive heart failure within 6 months before screening;
* Pregnant women, nursing mothers, or reluctant to agree taking effective contraceptive measures during the period of trial subjects;
* Those who have other neurological diseases or disabilities or mental diseases, which may affect the efficacy evaluation of this study as judged by the investigator;
* Those with a history of malignant tumor within 5 years before screening (if the patient has basal cell carcinoma of the skin or carcinoma in situ of the cervix and has been cured, he/she can participate in this study);
* Those who participated in other drug/device clinical studies and used the experimental drug/device within 3 months before screening;
* Any condition that, in the judgment of the investigator could impose hazards to the patient if study therapy is initiated or affect the participation of the patient in the study。

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Outcome | 90 days
  Proportion of subjects of excellent outcome defined as modified Rankin Scale (mRS) (0-1) at 90 days. mRS is a 7 grade scale from 0 to 6, where 0 is the best and 6 is the worst outcome.
Primary Safety Outcome | 90 days
  Proportion of patients with adverse events at 90 days.

SECONDARY OUTCOMES:
Infarction Volume | 14 days
  Infarction volume at 14 days compared to baseline
National Institutes of Health Stroke Scale (NIHSS) | 72 hours， 7 days， 14 days， 90days
  National Institutes of Health Stroke Scale (NIHSS) score changes from baseline. NIHSS is 42 point scale where 0 is the best o and 42 is the worst outcome.
Excellent functional outcome | 14 days
  Favourable outcome rate is defined as the proportion of subjects with modified Rankin Scale (mRS) (0-1). mRS is a 7 grade scale from 0 to 6, where 0 is the best and 6 is the worst outcome.
Modified Rankin Scale (mRS) distribution | 14 days， 90 days
  Ordinal distribution of Modified Rankin Scale (mRS). mRS is a 7 grade scale from 0 to 6, where 0 is the best and 6 is the worst outcome.
Barthel index (BI) | 90 days
  Proportion of subjects with Global function of daily living defined as Change in Barthel index (BI) ≥ 95. BI is a 10 item scale with scores ranging from 0 to 100, where a score of 100 is the best and 0 is the worst outcome.
Symptomatic intracranial hemorrhage(sICH) | 14 days
  Proportion of subjects with symptomatic intracranial hemorrhage (sICH)
AEs | 72 hours，7 days， 14 days
  Proportion of subjects with AEs
SAEs | 72 hours，7 days， 14 days，90days
  Proportion of subjects with SAEs

OTHER OUTCOMES:
Biomarkes | 14 days
  The changes of serum high sensitivity C-reactive protein test (hs-CRP) level from baseline to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, M.D., Principal Investigator — Beijing Tiantan Hospital, Capital Medical University, Beijing, China
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China